CLINICAL TRIAL: NCT06231173
Title: Effects of Visual Feedback Therapy on Post Burn Hand Contractures in Children
Brief Title: Effects of Visual Feedback Therapy on Post Burn Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0732
Record Dates: First submitted 2023-12-26; First posted 2024-01-30 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Burn Hand
Keywords: Burns, Goniometer, Hand contractures; Visual feedback therapy
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Visual feedback therapy and conventional therapy
  Interventions: Other: Visual Feedback Therapy and Conventional Therapy
- Controlled (Active Comparator): Conventional therapy
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Visual Feedback Therapy and Conventional Therapy — In experimental group individuals will receive visual feedback therapy and Conventional rehabilitation therapy. In visual feedback therapy, bilateral method is used to receive the visual feedback from the mirror. This visual feedback therapy consists of the following parts as the patient is asked to follow the involved hand that did the mimicking while the non-involved side will be performing wrist flexion, wrist extension, ulnar deviation, radial deviation, supination, pronation, and closing hand and opening hand.In conventional therapy, Patients are given a rest time of 20 seconds in each activity and a 1-minute break in each segment in order to reduce fatigue of the noninvolved hand. The treatment will be applied by the therapist standing at the side of the patient. Then technique will be applied according to subject's tolerance for duration of 15 minutes in each sitting. This treatment protocol will be 5 times/week for 4 weeks in the hospital setting.
  Arms: Experimental
Other: Conventional Therapy — In control group individuals will receive only conventional therapy. In conventional therapy, Patients are instructed to perform a sandbag and hand grip exercise with a resistive exercise for the non-involved side. At last, patients are instructed to perform a moving small object (ball of wool) and card flip operation to induce wrist and finger movements as functional activities. Patients are given a rest time of 20 seconds in each activity and a 1-minute break in each segment in order to reduce fatigue of the non involved hand. The treatment will be applied by the therapist standing at the side of the patient. Then technique will be applied according to subject's tolerance for duration of 15 minutes in each sitting. .This treatment protocol will be 5 times/week for 4 weeks in the hospital setting.
  Arms: Controlled

SUMMARY:
Visual feedback therapy is a cheap, easy, and, most importantly, patient-directed treatment that may improve the recovery of hand motor functional skills. Visual feedback therapy consists of repeated bilateral, symmetrical movements in which the patient moves the affected body part as much as he/she could while observing the reflection.The hands account for less than 5 % of total body surface area. Many burns requiring hospitalization involve the upper extremity considered severe injuries by the American Burn Association and should be referred to specialized care centers to minimize sequella of thermal injury including nail deformities, hypertrophic scars, boutonniere deformity, digit loss, and contractures. Visual feedback therapy is a treatment method based on neuroplasticity of the brain.Although recent studies have demonstrated the benefit of visual feedback therapy for various diseases, research that applies visual feedback therapy to improve the restorative capability of hand function of patients with reduced hand function due to mutilated injury has not been reported yet.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial. Study will be approved by ethical committee. After that informed consent will be taken and patients will be included in the study based on the inclusion criteria. Non probability convenience sampling technique will be used and study will be conducted on 36 patients diagnosed with post burn hand contractures 8-12 years old children. Patient will be randomly categorized into two groups by using flip coin method. Experimental group will receive visual feedback therapy and conventional therapy treatment protocol. Control group will receive only conventional therapy. Pre and Post interventions assessment will be made for both groups. Post burn hand contractures of the patients will be assessed by checking ROMS of hands with goniometer. The ABILHAND questionnaire will also be performed to check the functional movements of hands and visual analogue scale will be used for pain assessment. Data will be analyzed by using SPSS 25.0 statistical tool. Appropriate statistical test will be used after checking normality of data.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 12 years old children with post burn hand contractures
* Patients with flame burns
* Patients with 2nd degree burns

Exclusion Criteria:

* Patients with hand burns with any post burn complications
* Patients with wound infections
* Patients with 3rd degree burns Patients with hand fractures

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Goniometer | 4 weeks
  Goniometer both for upper and lower limb, is the simplest and most extended tool for measuring ROM in the clinical practice It was developed approximately 60 years ago, and its versatility and usability led to this instrument being promptly integrated into the field of physiotherapy and rehabilitation as a helpful evaluation tool. The intra-class correlation coefficients (ICC) ranged from 0.94 to 0.97 from the goniometric measurements
THE ABILHAND | 4 weeks
  The ABILHAND is a Rasch-based assessment that measures patients' perceived difficulty in performing ADLs that require the use of the bilateral upper limbs. It contains 23 items measuring manual ability and is rated on a 3-point response scale. The score, given in logits, is the conversion of the ordinal score into a linear measure of ability located on a unidimensional scale. The ABILHAND is a scale measuring bimanual ability that is often used to determine the level of UE dysfunction. Most of the validity studies on the ABILHAND demonstrated that the ABILHAND measured the concept of motor ability in a "standardized" or natural environment by significant correlations between the ABILHAND and grip strength, motricity, dexterity, or actual UE performance as measured by the accelerometers
Visual analogue scale (VAS) | 4 weeks
  Visual analogue scale (VAS) is a scale used for pain assessment, horizontal line 100mm in length, anchored by word descriptors at each end. The patient was asked to mark on the line the point they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks

CONTACTS AND LOCATIONS:
Overall Officials: Sana Mushtaq, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tofani M, Santecchia L, Conte A, Berardi A, Galeoto G, Sogos C, Petrarca M, Panuccio F, Castelli E. Effects of Mirror Neurons-Based Rehabilitation Techniques in Hand Injuries: A Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2022 May 2;19(9):5526. doi: 10.3390/ijerph19095526. PMID 35564920
- [Background] Wang TN, Lin KC, Wu CY, Chung CY, Pei YC, Teng YK. Validity, responsiveness, and clinically important difference of the ABILHAND questionnaire in patients with stroke. Arch Phys Med Rehabil. 2011 Jul;92(7):1086-91. doi: 10.1016/j.apmr.2011.01.020. PMID 21704789